CLINICAL TRIAL: NCT03960034
Title: Cachexia in Advanced NSCLC Patients: Diagnosis, Characterization, Prognosis, Functional Implications and Validation of Skeletal Muscle Disfunction Markers
Brief Title: Cachexia in NSCLC Patients: Diagnosis, Characterization, Prognosis, Functional and Skeletal Muscle Implications
Acronym: LUCAX01
Status: Completed | Type: Observational
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: NP802/15
Record Dates: First submitted 2019-04-18; First posted 2019-05-22 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: NSCLC Stage IV
Keywords: Cachexia; Skeletal Muscle Atrophy; Physical Functional Performance; Prognosis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Cachexia; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skeletal muscle from vastus lateralis and whole blood, blood plasma and peripheral blood mononuclear cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
LUCAX01 is a cohort study with patients with advanced NSCLC in tobacco users. in this study, patients will be submitted to baseline physical tests, blood and biopsy sample collection, and the main objective is to study the functional and prognostic implications of cachexia and to validate skeletal muscle dysfunction markers.

DETAILED DESCRIPTION:
Non-small-cell lung cancer (NSCLC) is currently the neoplasm leading in deaths worldwide and in Brazil, it figures as the second most common cancer in terms of the number of deaths. Patients are usually diagnosed in advanced stages and, consequently, more than 45% of all patients are diagnosed with cachexia. This syndrome is characterized by a loss of muscle mass with or without fat loss and it cannot be reversed by nutritional support. In the physiopathology of cachexia, generally are present exacerbated inflammation, severe loss of muscle contractile proteins, leading to fatigue and increased mortality. Furthermore, patients with cachexia usually do present lower response rates to anticancer treatments and it is also associated with a worse overall prognosis.

Treatments directed to mitigate muscle loss in these patients are awaited. Cohort studies do suggest a significant positive impact of physical fitness and prognosis in different chronic diseases; however, its impact in advanced NSCLC patients is not clear. Here our aim is to better understand the relationship between cachexia and physical fitness variables (muscle and cardiorespiratory function, body composition, and daily physical activity level) with prognosis and mortality in a group of NSCLC patients, as well as to study the effect of chemotherapy on these variables. Besides that, will be evaluated the skeletal muscle, Treg lymphocytes, and inflammatory biomarkers and compare cachectic and non-cachectic patients.

Sixty NSCLC patients will be accrued. Will be assessed the maximum oxygen consumption, daily physical activity, muscle function, muscle morphology, anxiety, depression, performance status, and fatigue pre-treatment. Blood and muscle biopsy samples will be collected. The prognostic impact of these physical fitness variables will be defined, as well as their predictive value in terms of response to anticancer treatments in advanced NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage IVa or IVb NSCLC patients histologically diagnosis.
* Eastern Cooperative Oncology Group Performance status 0 - 2
* Treatment-naive
* Current smokers or ex-smokers
* Normal renal, hepatic and hematological functions
* Able to perform the physical functional tests
* Able to read and sign the consent form

Exclusion Criteria:

* Initiate treatment before initiate
* Diagnostic of tumor mutation ( epidermal growth factor receptor, Anaplastic lymphoma kinase)

Obs: A smoker population with no known cancer will be used as controls (n=10)

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: NSCLC patient, current smokers or ex-smokers treatment naive with good Eastern Cooperative Oncology Group Performance status (ECOG-PS). A smoker population with no known cancer will be used as controls (n=10)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Overall survival in cachectic and non-cachectic patient | 2 year
  Survival will be measured to understand the prognostic impact of cancer cachexia in NSCLC patients.

SECONDARY OUTCOMES:
Physical fitness and response to treatment | 1 year
  Response Evaluation in solid tumors (RECIST 1.1) will be used to evaluate the relationship between physical fitness and response to chemotherapy.
Physical fitness and toxicity | 1 year
  Common terminology criteria for adverse events (CTCAE 5.0) will be used to evaluate the relationship between physical fitness and toxicities related to chemotherapy.
Cancer cachexia skeletal muscle pathways | 1 year
  Determination of down and up-regulated skeletal muscle pathways cachectic and non-cachectic patient using RNA-sec.
Cluster of Differentiation 4+ (CD4+) population in cachectic and non-cachectic patient. | 1 year
  Determination of CD4+ profile in cachectic and non-cachectic patients using flow cytometry.
Cluster of Differentiation 25+ (CD25+) population. | 1 year
  Determination of CD25+ profile in cachectic and non-cachectic patients using flow cytometry.
Forkhead box P3 regulatory T (Fox-p3+) population. | 1 year
  Determination of Fox-p3+ profile in cachectic and non-cachectic patients using flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto de Castro Junior, MD, PhD, Principal Investigator — Instituto do Câncer do Estado de São Paulo - FMUSP
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo, Brazil